CLINICAL TRIAL: NCT04210700
Title: Comparing Fascia Iliaca Compartment Block With Pericapsular Nerve Group Block for Hip Fracture Pain Control Before Operation
Brief Title: Comparing Fascia Iliaca Compartment Block and Pericapsular Nerve Group Block for Hip Fracture Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Chin Kao, Attending physician, Department of Anesthesiology, Principal investigator,, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19MMHIS254e
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Hip Fractures; Analgesia; Nerve Blocks
MeSH Terms: conditions — Hip Fractures; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia iliaca compartment block (Active Comparator): Participants will receive fascia iliaca compartment block before spinal anesthesia and operation
  Interventions: Procedure: Fascia iliaca compartment block
- Pericapsular nerve group block group (Experimental): Participants will receive pericapsular nerve group block before spinal anesthesia and operation
  Interventions: Procedure: Pericapsular nerve group block

INTERVENTIONS:
Procedure: Fascia iliaca compartment block — A linear ultrasound transducer is placed in a sagittal plane to identify the anterior superior iliac spine. By sliding the transducer medially, the fascia iliaca and abdominal internal oblique, sartorius, and iliopsoas muscles are identified. After identifying the "bow-tie sign", a 23-gauge needle (7mm, Nipro, Japan) is inserted in plane from caudal to cephalad until the needle tip penetrate the fascia iliaca. After negative aspiration, 0.35% ropivacaine 30mL with 1:400,000 epinephrine will be injected to separate the fascia iliaca and the iliacus muscle.
  Arms: Fascia iliaca compartment block
Procedure: Pericapsular nerve group block — A curvilinear ultrasound transducer is initially place on the anterior inferior iliac spine and then aligned to the iliopubic eminence by rotating around 45 degree. In this view, the iliopubic eminence, iliapsoas muscle and tendon, pectineus muscle, femoral artery and vein will be identified. A 23-gauge needle (7mm, Nipro, Japan) is inserted in plane from lateral to medial until the needle tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. After negative aspiration, 0.35% ropivacaine 20mL with 1:400,000 epinephrine will be injected.
  Arms: Pericapsular nerve group block group

SUMMARY:
The aim of the study is to compare the analgesic effect of fascia iliaca compartment block (FIC) block and pericapsular nerve group (PENG) block in hip fracture pain control. The participants, caregivers, and assessors will be blinded to the type of block the participants receive. Patients aged 20 years or older with hip fracture scheduled for surgical treatment will be assessed for eligibility to participate the study. One hundred eligible patients will be included in the study after informed consents are obtained, and then randomly allocated into either FIC block or PENG block, with 50 patients in each group. Both blocks will performed under ultrasound guidance.

The followings will be assessed: the numerical rating pain scale (NRS 0-10, 0: no pain, 10: worst pain imaginable) at before and after nerve block at different time points during rest and passive internal rotation of the fractured lower limb to neutral position from its typical external rotation deformity 30 mins after block (primary outcome). The degree of patient's satisfaction regarding nerve blocks and anesthesiologist's satisfaction regarding patient position during spinal anesthesia will also be assessed. The pain and use of rescue analgesics in the first 24 hours after operation will be recorded.

DETAILED DESCRIPTION:
The aim of this study is to compare the analgesic effect of fascia iliaca compartment block (FIC) block and pericapsular nerve group (PENG) block in hip fracture pain control before operation.

Methods This will be a randomized, assessor and participant-blinded study. After the patients give his /her informed consents, his/her baseline demographic data (gender, age, height, and body weight) and types of hip fracture will be recorded. Participants will be randomly allocated into either FIC block or PENG block by using the website RESEARCH RANDOMIZER (https://www.randomizer.org). One of the two anesthesiologists experienced in performed the FIC and PENG blocks will perform the nerve blocks. Only the anesthesiologist performing the nerve block and his assistant will be aware of which nerve block the participant receives immediately before performing nerve block by opening a sealed envelope. The assessors, in-charge anesthesiologists and nurse anesthetists, operation room personnel, surgeons and study participants will be all blinded to the randomization.

On arrival of the operating theater, all participants will be sent to the nerve block area, where continuous electrocardiogram, pulse oximetry, and non-invasive intermittent blood pressure monitoring will be applied and an intravenous line will be established. Before any intervention, pain at rest and during the fractured lower limb being passively internal rotated in extension to neutral position from its usual externally rotated deformity by assessors will assessed using NRS. If the participant cannot tolerate passive internal rotation of his/her fractured limb due to pain, impossibility to perform the test will be recorded as well as the worst NRS score during these attempts. The same assessment will be performed every 10 mins for until 30 mins after completion of the nerve block. Then the patient will be sent to the operation room, where spinal anesthesia will be performed for the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgical treatment for hip fracture
* American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* allergy to local anesthetics
* pregnancy
* inability to understand and use the numerical rating scale (NRS 0-10, 0: no pain, 10: worst pain imaginable) after instruction
* chronic use of opioids
* coagulopathy
* neuropathy
* severe diabetic mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-04 (Actual)

PRIMARY OUTCOMES:
Pain measurement at rest | 30 minutes after nerve blocks
  Numerical pain rating scale (0-10, 0: no pain, 10: worst pain imaginable) at rest
Pain measurement during internal rotation | 30 minutes after nerve blocks
  Numerical pain rating scale (0-10, 0: no pain, 10: worst pain imaginable) during the fractured limb being passively internally rotated to neutral position from usual externally rotated deformity

SECONDARY OUTCOMES:
Pain measurement at rest | 10 minutes after nerve block
  Numerical pain rating scale (0-10, 0: no pain, 10: worst pain imaginable) at rest
Pain measurement during internal rotation | 10 minutes after nerve block
  Numerical pain rating scale (0-10, 0: no pain, 10: worst pain imaginable) during the fractured limb being passively internally rotated to neutral position from usual externally rotated deformity
Pain measurement at rest | 20 minutes after nerve block
  Numerical pain rating scale (0-10, 0: no pain, 10: worst pain imaginable) at rest
Pain measurement during internal rotation | 20 minutes after nerve block
  Numerical pain rating scale (0-10, 0: no pain, 10: worst pain imaginable) during the fractured limb being passively internally rotated to neutral position from usual externally rotated deformity
pain measurement during positioning for spinal anesthesia | Just before operation
  Numerical pain rating scale (0-10, 0: no pain, 10: worst pain imaginable) during changing position from supine to lateral decubitus with flexion of the healthy hip
pain measurement after operation | 6, 12, and 24 hours after operation
  Numerical pain rating scale (0-10, 0: no pain, 10: worst pain imaginable)
the time spending for performing spinal anesthesia | Just before operation
  defined as starting of positioning maneuver to removal of spinal needle
quality of position for spinal anesthesia | Just before operation
  characterized as unsatisfied, satisfied, good, and excellent by the anesthesiologists performing the spinal anesthesia
the first time of pain perceived by the patient after operation | Within 48 hours after operation
  the time interval between the end of operation and pain first perceived by the patient
the time of first request for rescue analgesics after operation | Within 48 hours after operation
  the time interval between the end of operation and the first request for rescue analgesics
total consumption of rescue analgesics within 24 hours after the operation | Within 24 hours after the operation
  total consumption of rescue analgesics within 24 hours after the operation
the first time of ambulation after operation | Within 72 hours after operation
  the time interval between the end of operation and the first time the patient can ambulate with assistance after operation
the time spending for nerve block | Before operation
  defined as from contact of skin by the ultrasound transducer to removal of the needle

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chin Kao, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnell O, Kanis JA. An estimate of the worldwide prevalence and disability associated with osteoporotic fractures. Osteoporos Int. 2006 Dec;17(12):1726-33. doi: 10.1007/s00198-006-0172-4. Epub 2006 Sep 16. PMID 16983459
- [Background] Cooper C, Campion G, Melton LJ 3rd. Hip fractures in the elderly: a world-wide projection. Osteoporos Int. 1992 Nov;2(6):285-9. doi: 10.1007/BF01623184. PMID 1421796
- [Background] Bhandari M, Swiontkowski M. Management of Acute Hip Fracture. N Engl J Med. 2017 Nov 23;377(21):2053-2062. doi: 10.1056/NEJMcp1611090. No abstract available. PMID 29166235
- [Background] Beaudoin FL, Haran JP, Liebmann O. A comparison of ultrasound-guided three-in-one femoral nerve block versus parenteral opioids alone for analgesia in emergency department patients with hip fractures: a randomized controlled trial. Acad Emerg Med. 2013 Jun;20(6):584-91. doi: 10.1111/acem.12154. PMID 23758305
- [Background] Diakomi M, Papaioannou M, Mela A, Kouskouni E, Makris A. Preoperative fascia iliaca compartment block for positioning patients with hip fractures for central nervous blockade: a randomized trial. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):394-8. doi: 10.1097/AAP.0000000000000133. PMID 25068412
- [Background] Steenberg J, Moller AM. Systematic review of the effects of fascia iliaca compartment block on hip fracture patients before operation. Br J Anaesth. 2018 Jun;120(6):1368-1380. doi: 10.1016/j.bja.2017.12.042. Epub 2018 Apr 5. PMID 29793602
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Desmet M, Vermeylen K, Van Herreweghe I, Carlier L, Soetens F, Lambrecht S, Croes K, Pottel H, Van de Velde M. A Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty. Reg Anesth Pain Med. 2017 May/Jun;42(3):327-333. doi: 10.1097/AAP.0000000000000543. PMID 28059869
- [Background] Vermeylen K, Desmet M, Leunen I, Soetens F, Neyrinck A, Carens D, Caerts B, Seynaeve P, Hadzic A, Van de Velde M. Supra-inguinal injection for fascia iliaca compartment block results in more consistent spread towards the lumbar plexus than an infra-inguinal injection: a volunteer study. Reg Anesth Pain Med. 2019 Feb 22:rapm-2018-100092. doi: 10.1136/rapm-2018-100092. Online ahead of print. PMID 30798268
- [Background] Candal-Couto JJ, McVie JL, Haslam N, Innes AR, Rushmer J. Pre-operative analgesia for patients with femoral neck fractures using a modified fascia iliaca block technique. Injury. 2005 Apr;36(4):505-10. doi: 10.1016/j.injury.2004.10.015. PMID 15755432

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT04210700/Prot_SAP_000.pdf